CLINICAL TRIAL: NCT05370846
Title: The Impact of the Establishment of a New Antimicrobial Stewardship (AMS) Clinical Pharmacy Service in a Rural Hospital in Austria
Brief Title: The Impact of the Establishment of a New AMS CPS in a Rural Hospital in Austria
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Ulster (Other)
Collaborators: Northern Health and Social Care Trust (Other Government); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Aaron Courtenay, Lecturer in Clinical Pharmacy, University of Ulster
Other Study IDs: 437717
Record Dates: First submitted 2022-03-28; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Antimicrobial Stewardship

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical pharmacy antimicrobial stewardship intervention — A new AMS group will be introduced in Tauernklinikum in Zell am See, based on the S3-AWMF-guideline "Strategien zur Sicherung rationale Antibiotika-Anwendung im Krankenhaus" on antibiotic use in hospitals. As part of this, a new formulary will be developed and gradually introduced where we determined which AMS guidelines need to be incorporated. Antimicrobial use will be audited after set-up of the local formulary against the data from before implementation (using defined daily dose, DDD, as suggested by the WHO). Data on antimicrobial use will be obtained from a recently purchased and installed AMS programme called HyBase® by epiNET AG. AMS group will be provided with implementation material and toolkits, baseline data for antimicrobial use within hospital will be obtained.

SUMMARY:
Antimicrobial stewardship groups ensure the safe and prudent use of antibiotics, decrease antimicrobial resistance, lower costs of antimicrobials in hospital settings and improve patient safety in terms of prescribing plausibility. Significant success of the implementation of antimicrobial stewardship programmes have been shown in studies across the world. It is important to highlight this issue not only because of the current alarming resistance situation but also to encourage Austrian stakeholders and politicians to start to implement such programmes on a larger scale all across Austria.

DETAILED DESCRIPTION:
Antimicrobial stewardship groups ensure the safe and prudent use of antibiotics, decrease antimicrobial resistance, lower costs of antimicrobials in hospital settings and improve patient safety in terms of prescribing appropriateness. Significant success following the implementation of antimicrobial stewardship programmes have been shown in studies across the world. It is important to highlight this issue not only because of the current alarming antimicrobial resistance situation but also to encourage Austrian and European stakeholders and politicians to start to implement such programmes on a larger scale across Austria. There are AMS groups in place in larger Austrian healthcare facilities. However, in Austria only 15.3% of all hospitals have a hospital pharmacy and only a small part of them offer clinical pharmacy services (CPS). Clinical pharmacy projects need to be put into place demonstrating the positive impacts for both patients and the healthcare system and the data published to make the advantages publicly available and visible in order to achieve legal changes in Europe. A hospital pharmacy should be a requirement in every hospital and the delivery of CPS should be compulsory. AMS is a well-known expertise in anglophone countries, and this is a great opportunity to demonstrate the importance and need for such a service in all European countries. Setting up AMS groups should be statutory in order to raise awareness of and to combat antimicrobial resistance. Globally speaking, if more small hospitals focus on developing AMS strategies, then it will be possible to deliver the requirements of both the WHO global action plan and the European Commission's "A European One Health Action Plan against Antimicrobial Resistance (AMR)" to optimize the use of antimicrobials in humans.

This will be a very valuable project for Austria as it is a collaboration between Tauernklinikum in Zell am See, Antrim Hospital in Northern Ireland, the Medicines Optimization Innovation Centre (MOIC) and Ulster University. The United Kingdom has been the distinct European leader of clinical pharmacy services (CPS) implementation with an AMS group setup being one of their specialties. The MOIC has pioneered work in many CPS fields and with the support and guidance of MOIC, Antrim hospital and Ulster University as leading institutions for CPS in Europe this project will be a success. It will not only promote AMS across Europe but also strengthen and develop the clinical pharmacy profession. MOIC is currently involved with work in this area in both Poland and Estonia, which will further enable synergies and sharing and learning with this project much more widely.

A new AMS group will be introduced in Tauernklinikum in Zell am See, based on the S3-AWMF-guideline "Strategien zur Sicherung rationale Antibiotika-Anwendung im Krankenhaus" on antibiotic use in hospitals. As part of this, a new formulary will be developed and gradually introduced where we determined which AMS guidelines need to be incorporated. Antimicrobial use will be audited after set-up of the local formulary against the data from before implementation (using defined daily dose, DDD, as suggested by the WHO). Data on antimicrobial use will be obtained from a recently purchased and installed AMS programme called HyBase® by epiNET AG. AMS group will be provided with implementation material and toolkits, baseline data for antimicrobial use within hospital will be obtained.

Data will be collated prior to implementation of the AMS group and after the group has been established (3 months after antimicrobial ward rounds implementation - planned Q4 this year and over the following two years), when it will be compared to the agreed guidelines. Evaluation of this data will determine the impact of the group's activities on prescribing generally and adherence to guidelines specifically.

The AMS group should help ensure effective collaboration between the various members of the healthcare team in the hospital and allow employees to attend relevant training courses or hear educational talks on site. The whole process will raise awareness, improve patient outcomes and prescribing habits and reduce hospital costs. A special focus will be put on enhancing the liaison between laboratory, IT, pharmacy, care personnel and medical staff. Prescribers should be able to rely on their own skills but also collaborate with other professionals' thereby also maximizing their competencies.

Anecdotal evidence suggests that it is difficult to make AMS work when multidisciplinary collaboration is not established. The study site size of a small 350 bed hospital is perfect to analyze the improvement of multiprofessional cooperation in this process. The AMS group will be set up including staff from nursing, medical, pharmacy, laboratory and IT. The effectiveness of the group will be evaluated for via questionnaire and focus groups in the individual departments at the implementation of the ward rounds and again one year later. The patient perspective of the service will also be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients of Tauernklinikum in Zell am See receiving antimicrobial treatment between 13th April 2022 and 12 April 2025

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients from all wards will be included in this study, all adult and paediatric patients will be included. Interpreting services will be available as required.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-05-09 (Estimated); Primary Completion 2025-04-12 (Estimated); Study Completion 2025-04-12 (Estimated)

PRIMARY OUTCOMES:
Identifying risk factors for inappropriate antimicrobial prescribing across prescribers and regions and improvement strategies | 3 years
  Risk factors for inappropriate prescribing will be determined via using medication appropriateness index (MAI), de-escalation rates and hospital length of stay (considering reduction of bed days both measured in number of days).
Identifying risk factors for ineffective antimicrobial prescribing across prescribers and regions and improvement strategies | 3 years
  Ineffective antimicrobial prescribing will be addressed as per antibiotic consumption (defined daily doses DDD, antimicrobial therapy duration in numbers of days), patient bed days in numbers of days and readmission rates within six months of last inpatient stay.
Cost change of effective antibiotic prescribing | 3 years
  Cost change of effective antibiotic prescribing will be measured in Euros.

SECONDARY OUTCOMES:
Impact of AMS interventions on outcomes | 3 years
  A new antimicrobial formulary will be implemented and prescribing habits will be assessed against it after implementation. This will be done via data extracted from HyBase anti-infective surveillance software and auditing electronic patient cardexes. As suggested by the WHO DDD defined daily doses will be utilised.
Cost-consequence analysis | 3 years
  Cost-consequence analysis will be performed for the implementation of new AMS interventions and the introduction of a new antimicrobial hospital formulary.
Assessment of patient's Quality of life (QoL) | 3 years
  The number of hospital bed days (length of stay) will be recorded
Introduction of antimicrobial surveillance software system | 3 years
  HyBase software will be introduced which will capture the frequency of "alert" organisms.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Courtenay, Dr., Principal Investigator — PI of the study

IPD SHARING:
Plan to Share IPD: No
Fully anonymised data only will be shared with the wider research team.